CLINICAL TRIAL: NCT02234271
Title: Plan A Birth Control: Randomized Controlled Trial of a Mobile Health Application for Contraception Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, UCLA Women's Health Clinical Research Unit, Department of Obstetrics and Gynecology, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: UCLA_IRB_14-000821
Record Dates: First submitted 2014-08-26; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Mobile Applications; Contraception; Contraception Behavior
MeSH Terms: conditions — Contraception Behavior

ARMS (2):
- Health Educator Arm (Active Comparator): Health Educator for contraception information
  Interventions: Other: Health Educator Counseling
- Mobile Health Application Arm (Experimental): Plan A Birth Control - iPad based application for contraception information
  Interventions: Other: Mobile Health Application

INTERVENTIONS:
Other: Mobile Health Application — Mobile Health application for contraception information
  Arms: Mobile Health Application Arm
Other: Health Educator Counseling — Counseling via health educator
  Arms: Health Educator Arm

SUMMARY:
The primary objective of the investigators study was to design a comprehensive and medically accurate contraception counseling mobile health application and evaluate the effects of this contraception counseling application on the contraceptive methods that patients selected and their knowledge of that method.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* literate in English
* not at that time using a contraceptive method
* willing to switch to a new reversible contraceptive method
* currently sexually active with a male partner and
* intending to avoid pregnancy for at least one year

Exclusion Criteria:

* women not at risk for unintended pregnancy
* those who were pregnant
* seeking pregnancy within the next 12 months
* history of surgical sterilization or
* a current partner who had had a vasectomy
* using long acting reversible birth control method
* menopausal

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Contraception choice | Participants were followed for the duration of their clinic visit which was up to one day
  Choice of birth control selected by participant was recorded into electronic database system and compared between the two groups.

SECONDARY OUTCOMES:
Knowledge of contraception method chosen | Participants were followed for the duration of their clinic visit which was up to one day
  A knowledge questionnaire was administered at the end of patient's visit and results were analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Sridhar, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- West Medical Clinic, Los Angeles, California, United States

REFERENCES:
- [Derived] Sridhar A, Chen A, Forbes ER, Glik D. Mobile application for information on reversible contraception: a randomized controlled trial. Am J Obstet Gynecol. 2015 Jun;212(6):774.e1-7. doi: 10.1016/j.ajog.2015.01.011. Epub 2015 Jan 9. PMID 25582097